CLINICAL TRIAL: NCT01579851
Title: Recovery After Sugammadex(TIVA Using Propofol vs Inhalation Anesthesia Using Sevoflurane)
Brief Title: Recovery After Sugammadex(Propofol vs Sevoflurane)
Acronym: Sugammadex2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/58; 2010-023943-13 (EudraCT Number)
Record Dates: First submitted 2012-01-04; First posted 2012-04-18 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Anesthesia
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol-Remifentanil (Active Comparator): Anesthesia is maintained with Propofol and Remifentanil; myorelaxation is obtained with rocuronium
  Interventions: Drug: Sugammadex
- Sevoflurane-Remifentanil (Active Comparator): Anesthesia is maintained with Sevoflurane and Remifentanil; myorelaxation is obtained with rocuronium
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — sugammadex
  * 4 mg/kg : if there is no response to Train of Four stimulations and at least one response to the Post Tetanic Count
  * 2 mg/kg : if there is at least two responses to Train of Four stimulations

SUMMARY:
Sugammadex is used to reverse of a neuro-muscular block deep. It has been reported that its administration could induce signs of recovery despite continuation of anesthetic drugs. The goal of the present study is to look is the arte of this event is different according to the primary anesthetic agent used.

ELIGIBILITY:
Inclusion Criteria:

* adult patients scheduled to receive general anesthesia with muscle relaxation achieved with rocuronium

Exclusion Criteria:

* Known drug allergy,
* Contra-indications to the use of propofol, remifentanil, rocuronium, sevoflurane, sugammadex
* Difficulty to use Bispectral Index monitor
* Inability to obtain a proper monitoring of muscle relaxation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with an increase in Bispectral Index after sugammadex injection | One hour after anesthesia
  Increase in Bispectral Index (> 20) after sugammadex injection
Number of patients with occurence of clinical signs of awakening after sugammadex injection | One hour after anesthesia
  Clinical signs of awakening after sugammadex are wallowing, eye opening on demand, cough, spontaneous movements, response to simple commands, tearing, ...

SECONDARY OUTCOMES:
T4/T1 ratio after sugammadex injection | One hour after anesthesia
  Modification of T4/T1 ratio after sugammadex injection
Number of patients with side effects due to sugammadex injection | One hour after anesthesia
  Side effects after sugammadex injection are bradycardia, nausea or vomiting, pain, residual curarisation, awareness,...

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Le Guen, MD, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, Île-de-France Region, France